CLINICAL TRIAL: NCT01523808
Title: Phase I, Dose Escalation Clinical Trial of GRASPA (Red Blood Cells Encapsulating L-Asparaginase) in Patients With Pancreatic Carcinoma
Brief Title: Administration of GRASPA (Suspension of Erythrocytes Encapsulating L-asparaginase)in Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ERYtech Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRASPANC2008-02
Record Dates: First submitted 2012-01-16; First posted 2012-02-01 (Estimated); Results first posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-08

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; asparaginase
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- GRASPA 25 (Experimental)
  Interventions: Drug: GRASPA
- GRASPA 50 (Experimental)
  Interventions: Drug: GRASPA
- GRASPA 100 (Experimental)
  Interventions: Drug: GRASPA
- GRASPA 150 (Experimental)
  Interventions: Drug: GRASPA

INTERVENTIONS:
Drug: GRASPA — Each patient will receive one administration of GRASPA . A stepwise increase of 4 single doses of GRASPA will be administered to cohorts of 3 patients per dose

SUMMARY:
The interest in using L-asparaginase in pancreatic cancer arose from in vitro and in vivo studies data showing an anti-neoplastic effect on pancreatic tumor cell lines. Interestingly, these studies suggest an additional effect of L-asparaginase associated to gemcitabine.GRASPA is a suspension of red blood cells encapsulating L-asparaginase. The aim of this phase I clinical trial is to evaluate the Maximum Tolerated Dose (MTD) of GRASPA on locally advanced or metastatic pancreatic tumors, after therapy failure of first or second line chemotherapy using gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* Exocrine pancreatic adenocarcinoma cytologically or histologically confirmed
* Locally advanced and non-resectable with invasion of the superior mesenteric artery (stage III) or metastatic (stage IV) as defined by TNM (primary tumor, regional nodes, metastasis) 2002 classification (UICC 2002)
* resistant to a first or second line chemotherapy with gemcitabine
* Patient aged between 18 to 70 years
* Signed Informed Consent Form
* Life expectancy ≥ 12 weeks
* Accurate measurement of tumor volume by imagery (in at least one dimension)
* Presence of one or several tumor markers (carcinoembryonic antigen [CEA] and cancer antigen [CA] 19.9)
* Eastern Cooperative Oncology Group [ECOG] Prognostic Score : 0, 1 or 2
* Patient beneficiary of a Social Security Insurance

Exclusion Criteria:

* Patient with an endocrine or acinar pancreatic tumor
* Patient with known or suspected cerebro-meningeal metastases
* Haemoglobin level greater than 13 g/L
* Patient hypersensitive to L-asparaginase or have had prior exposure to any form of L-asparaginase
* Splenic vein thrombosis < 3 months or under active treatment
* Anti-vitamin K treatment
* Hepatic Insufficiency unrelated to pancreatic cancer
* Renal insufficiency unrelated to pancreatic cancer
* Pancreatitis or pancreatitis history unrelated to pancreatic cancer
* Insulin-dependant diabetes mellitus unrelated to pancreatic cancer
* Current or prior coagulopathy disorders unrelated to pancreatic cancer
* ECOG Prognostic Score 3 or 4
* History of grade 3 blood transfusion reaction (life threatening situation)
* Presence of rare and dangerous anti-erythrocyte antibodies preventing from getting a compatible packed Red Blood Cells for the patient
* Patient already included in another clinical trial
* Pregnancy, breast-feeding or absence of secured contraception
* Unwillingness to sign the informed consent form

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

REFERENCES:
- [Derived] Bachet JB, Gay F, Marechal R, Galais MP, Adenis A, MsC DS, Cros J, Demetter P, Svrcek M, Bardier-Dupas A, Emile JF, Hammel P, Ebenezer C, Berlier W, Godfrin Y, Andre T. Asparagine Synthetase Expression and Phase I Study With L-Asparaginase Encapsulated in Red Blood Cells in Patients With Pancreatic Adenocarcinoma. Pancreas. 2015 Oct;44(7):1141-7. doi: 10.1097/MPA.0000000000000394. PMID 26355551

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 3 investigational sites in France between November 2009 and February 2011. The first participant was enrolled in the study on 27 November 2009 and the last patient exited the study on 30 March 2011.
Pre-assignment Details: This was not a randomized study. No washout or run-in was required. Assignment of patients to treatment groups followed study design rules, per protocol.
Period: Overall Study
Arm/Group | GRASPA 25 | GRASPA 50 | GRASPA 100 | GRASPA 150
Started | 3 | 3 | 3 | 3
Completed | 0 | 3 | 1 | 0
Not Completed | 3 | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- GRASPA 25: Participants received one administration of GRASPA . A stepwise increase of 4 single doses of GRASPA was administered to cohorts of 3 patients per dose
  3 subjects enrolled; 0 subjects completed
- GRASPA 50: Each patient will receive one administration of GRASPA . A stepwise increase of 4 single doses of GRASPA was administered to cohorts of 3 patients per dose
  3 subjects enrolled; 3 subjects completed
- GRASPA 100: Each patient will receive one administration of GRASPA . A stepwise increase of 4 single doses of GRASPA was administered to cohorts of 3 patients per dose
  3 subjects enrolled; 1 subject completed
- GRASPA 150: Each patient will receive one administration of GRASPA . A stepwise increase of 4 single doses of GRASPA was administered to cohorts of 3 patients per dose
  3 subjects enrolled; 0 subjects completed
- Total: Total of all reporting groups
Arm/Group | GRASPA 25 | GRASPA 50 | GRASPA 100 | GRASPA 150 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 3 | 1 | 8
  >=65 years | 0 | 2 | 0 | 2 | 4
Age, Continuous [Median (Full Range); unit: years] | 56 [55 to 59] | 67 [58 to 71] | 51 [43 to 62] | 68 [63 to 72] | 60 [43 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 1 | 3
  Male | 3 | 2 | 2 | 2 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  France | 3 | 3 | 3 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose-limiting Toxicities up to Week 4 After Treatment
Description: Dose limiting toxicities were defined according to CTCAE v3.0 as follow:
  Known toxicities related to asparaginase:
  * Pancreatic grade 2, 3 or 4
  * Allergic, Neurological, Hepatic, Coagulation grade 3 or 4 an any other toxicity of grade 4
Time Frame: 4 weeks
Measure: Number; unit: participants
Groups:
- GRASPA 25; GRASPA 150: GRASPA: Each patient will receive one administration of GRASPA . A stepwise increase of 4 single doses of GRASPA will be administered to cohorts of 3 patients per dose
  3 subjects enrolled; 0 subjects completed
- GRASPA 50: GRASPA: Each patient will receive one administration of GRASPA . A stepwise increase of 4 single doses of GRASPA will be administered to cohorts of 3 patients per dose
  3 subjects enrolled; 3 subjects completed
- GRASPA 100: GRASPA: Each patient will receive one administration of GRASPA . A stepwise increase of 4 single doses of GRASPA will be administered to cohorts of 3 patients per dose
  3 subjects enrolled; 1 subject completed
Arm/Group | GRASPA 25 | GRASPA 50 | GRASPA 100 | GRASPA 150
Number analyzed (Participants) | 3 | 3 | 3 | 3
participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Patients With Limiting Toxicities From Week 4 to Week 8 (End of Study)
Description: Limiting toxicities were defined according to CTCAE v3.0 as follow:
  Known toxicities related to asparaginase:
  * Pancreatic grade 2, 3 or 4
  * Allergic, Neurological, Hepatic, Coagulation grade 3 or 4 Any other toxicity of grade 4
Time Frame: 8 weeks
Population: AEs that met the following criteria were considered for the primary safety criterion:
  1. Grade 2 to 4 of pancreatic toxicity - no symptomatic pancreatitis occurred for any patients
  2. Grade 3 or 4 of hepatic toxicity - Two patients had antithrombin III decrease, but both cases were Grade 1; no cytolytic hepatitis
  3. Other grade 4 toxicities
Measure: Count of Participants; unit: Participants
Arm/Group | GRASPA 25 | GRASPA 50 | GRASPA 100 | GRASPA 150
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Encapsulated L-asparaginase Pharmacokinetic Parameters Terminal Half-life
Description: Pharmacokinetic (PK) parameters were analyzed for encapsulated asparaginase concentration data using Phoenix® WinNonlin® 6.3.
  Free and total L-asparaginase activity was measured during the study and encapsulated asparaginase was defined as the difference between total asparaginase and plasmatic asparaginase.
Time Frame: Days 0, 1, 3, 7, 14, 21, 28, 35, 42, 56
Population: Data were available for dose levels (no. of patients) of 25 IU/kg (n=1), 50 IU/kg (n=0), 100 IU/kg (n=0), and 150 IU/kg (n=3).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | GRASPA 25 | GRASPA 150
Number analyzed (Participants) | 1 | 3
days | 19.34 | 22.71 (10.48)

4. Secondary Outcome: Encapsulated L-asparaginase Pharmacokinetic Parameters Cmax
Description: as for outcome 3
Time Frame: Days 0, 1, 3, 7, 14, 21, 28, 35, 42, 56
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GRASPA 25 | GRASPA 150
Number analyzed (Participants) | 1 | 3
IU/L | 255.33 | 1812.57 (203.12)

5. Secondary Outcome: Encapsulated L-asparaginase Pharmacokinetic Parameters Area Under the Curve to Infinity
Description: as for outcome 3
Time Frame: Days 0, 1, 3, 7, 14, 21, 28, 35, 42, 56
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*IU/L
Arm/Group | GRASPA 25 | GRASPA 150
Number analyzed (Participants) | 1 | 3
hr*IU/L | 189363.84 | 1331430.20 (258279.50)

6. Secondary Outcome: Change of Asparagine Levels From Baseline (Pharmacodynamics)
Description: Duration of plasma asparagine depletion (less than or equal to 2 micromoles/Liter or deamination greater than 90% compared to baseline levels and serum concentrations of L-asparagine, L-aspartate, L-glutamine, and L-glutamate. For pharmacodynamic data, the administration date of the investigational treatment was considered as the reference date for duration calculation. All patients having received a single dose of studied drug GRASPA have been analyzed.
Time Frame: Days 0, 1, 3, 7, 14, 21, 28, 35, 42, 56
Population: 12 patients were included and analyzed corresponding to 1 cohort of 3 patients per dose. Data shown is a summary of the relative change of asparagine (%) from baseline over time (analysis set)
Measure: Mean (Standard Deviation); unit: UI/Kg
Arm/Group | GRASPA 25 | GRASPA 50 | GRASPA 100 | GRASPA 150
Number analyzed (Participants) | 3 | 3 | 3 | 3
UI/Kg
  Day 0 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Day 1: number analyzed (Participants) | 3 | 3 | 3 | 2
  Day 1 | -98.10 (0.35) | -98.36 (0.60) | -80.22 (31.67) | -97.26 (0.02)
  Day 3 | -98.10 (0.35) | -91.39 (11.49) | -72.66 (44.77) | -97.36 (0.18)
  Day 7 | -37.65 (55.53) | -80.06 (15.68) | -49.97 (52.19) | -93.02 (7.35)
  Day 14 | 3.74 (33.84) | -30.13 (11.06) | -6.63 (8.46) | -65.91 (54.30)
  Day 21 | 1.46 (52.13) | -13.21 (41.76) | -12.93 (9.87) | -31.64 (41.65)
  Day 28 | 8.77 (63.51) | -16.24 (40.46) | 0.94 (2.65) | -6.55 (8.54)
  Day 35: number analyzed (Participants) | 2 | 2 | 1 | 1
  Day 35 | -15.61 (33.87) | -10.95 (18.03) | 7.50 | 43.08
  Day 42: number analyzed (Participants) | 0 | 2 | 1 | 1
  Day 42 |  | -22.04 (47.31) | -7.81 | -1.82
  Day 56: number analyzed (Participants) | 0 | 1 | 1 | 0
  Day 56 |  | -74.80 | -7.26 |

7. Secondary Outcome: Number of Patient Positive for Anti-L-asparaginase Antibodies
Description: Titers of E. coli anti-asparaginase antibodies evaluated over time to assess immunogenicity
Time Frame: Day 0, 1, 28 and 56
Population: Summary of anti-L-asparaginase antibodies over time by number of patients
Measure: Count of Participants; unit: Participants
Arm/Group | GRASPA 25 | GRASPA 50 | GRASPA 100 | GRASPA 150
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants
  Day 0 | 0 | 0 | 1 | 0
  Day 1 | 0 | 0 | 0 | 0
  Day 28: number analyzed (Participants) | 3 | 3 | 3 | 2
  Day 28 | 2 | 3 | 3 | 0
  Day 56: number analyzed (Participants) | 0 | 2 | 1 | 2
  Day 56 |  | 2 | 1 | 2

8. Secondary Outcome: Summary of CEA Level Over Time
Description: Assess tumor response, evaluated by carcinoembryonic antigen (CEA) tumor marker evolution
Time Frame: Day 0, 28, 56
Population: Sample collection not completed at each timepoint for each patient. All data available presented below.
Measure: Median (Full Range); unit: ng/ml
Arm/Group | GRASPA 25 | GRASPA 50 | GRASPA 100 | GRASPA 150
Number analyzed (Participants) | 3 | 3 | 3 | 3
ng/ml
  Day 0: number analyzed (Participants) | 2 | 3 | 2 | 3
  Day 0 | 21.3 [13.5 to 29.0] | 10.2 [10.0 to 19.0] | 6.4 [3.0 to 9.7] | 354.8 [12.5 to 488.2]
  Day 28: number analyzed (Participants) | 2 | 3 | 2 | 3
  Day 28 | 22.8 [7.5 to 38.0] | 26.3 [7.5 to 30.9] | 3.1 [3.0 to 3.1] | 967.9 [14.2 to 995.4]
  Day 56: number analyzed (Participants) | 0 | 1 | 1 | 0
  Day 56 |  | 9.0 [9.0 to 9.0] | 3.4 [3.4 to 3.4] |

9. Secondary Outcome: Summary of CA 19.9 Over Time
Description: Tumor response Evaluation by cancer antigen (CA)19.9 evolution over time
Time Frame: Day 0, 28 and 56
Population: Sample collection not completed at each timepoint for each patient. All data available presented below.
Measure: Median (Full Range); unit: u/ml
Arm/Group | GRASPA 25 | GRASPA 50 | GRASPA 100 | GRASPA 150
Number analyzed (Participants) | 3 | 3 | 3 | 3
u/ml
  Day 0 | 18440.0 [5605.0 to 36802.0] | 184.3 [59.8 to 4751.0] | 1625.0 [73.2 to 2835.0] | 54.5 [3.5 to 1784.0]
  Day 28: number analyzed (Participants) | 2 | 3 | 2 | 3
  Day 28 | 37196.5 [14310.0 to 60083] | 748.3 [187.2 to 12375.0] | 3136.0 [122.0 to 6150.0] | 124.1 [5.3 to 2395.0]
  Day 56: number analyzed (Participants) | 0 | 1 | 1 | 0
  Day 56 |  | 561.8 [561.8 to 561.8] | 195.5 [195.5 to 195.5] |

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events starting from patient inclusion until 2 month after GRASPA administration (~2.5 months)
Description: Adverse events regardless of grade or causality are reported. Events are summarized by system organ class and footnote indicates the specific events reported for each class.
Arm/Group | GRASPA 25 | GRASPA 50 | GRASPA 100 | GRASPA 150
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/3 | 1/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 3/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 2/3 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GRASPA 25 (N=3) | GRASPA 50 (N=3) | GRASPA 100 (N=3) | GRASPA 150 (N=3)
Dyspnea related to pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Increase of Lumbar Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Increase of Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GRASPA 25 (N=3) | GRASPA 50 (N=3) | GRASPA 100 (N=3) | GRASPA 150 (N=3)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Diarrohea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gastroesophageal reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Astenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (3) | 1 (1) | 0 (0)
ECOG Performance Status worsened (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Antithrombin III decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No